CLINICAL TRIAL: NCT05576870
Title: Growth Study Using a Toddler Almond Based Nutritional Drink (Test) vs. a. Formula That Has Been Shown to Support Growth (Control) in Healthy Toddlers
Brief Title: Growth Study Using Else Toddler Nutritional Drink vs. a. Dairy Based Toddler Drink (Control) in Healthy Toddlers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Else Nutrition GH Ltd (Industry)
Collaborators: Children's Hosptial of Colorado Aurora, Colorado, United States (Unknown); Laina VTMS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Else001
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Weight Gain
Keywords: toddler; growth; nutrition
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant based toddler nutrition (Experimental): Plant based toddler nutrition based on almond and buckwheat drink
  Interventions: Other: Plant based toddler nutrition
- Dairy based toddler nutrition (Active Comparator): Commercially available dairy based toddler nutrition drink
  Interventions: Dietary Supplement: Dairy based toddler nutrition

INTERVENTIONS:
Other: Plant based toddler nutrition — Plant based toddler nutrition fed daily ad libitum
  Arms: Plant based toddler nutrition
Dietary Supplement: Dairy based toddler nutrition — Commercially available toddler nutrition fed daily ad libitum
  Arms: Dairy based toddler nutrition

SUMMARY:
The aim of the study is to investigate the growth of healthy toddlers fed with Toddler almond based nutritional drink (test) vs. a. formula that has been shown to support growth (control) in Healthy Toddlers

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age between ≥37 weeks + 0 days and ≤41 weeks + 6 days,
2. Weight for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
3. Length for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
4. Weight for length for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
5. Consuming and tolerating a cow's milk and almond at time of enrollment (at least 3 age appropriate portions)
6. Consuming and tolerating almond on more than one occasion in age appropriated doses, to ensure no reaction to study formula e.g. 2 teaspoons almond butter in one portion or 500 ml/16 fl oz per day

Exclusion Criteria:

1. Toddler with any positive food allergy test food allergy or intolerance to any foods
2. Participants are under ongoing medical care of a pediatrician which according to the parents will make it difficult to complete the study

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Weight gain | 4 months
height velocity | 4 months

SECONDARY OUTCOMES:
Daily intake | 4 months
  Volume of consumption will be recorded in fluid oz or ml per day

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided